CLINICAL TRIAL: NCT06141733
Title: 2 Year Follow up of COSGOD III (COSGOD III-FU)- Ancillary Retrospective Observational Study to COSGOD III Trial
Brief Title: 2 Year Follow up of COSGOD III
Acronym: COSGODIII-FU
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other); Medical University of Vienna (Other); Vittore Buzzi Children's Hospital (Other); University Hospital Tuebingen (Other); University College Cork (Other); University Hospital Freiburg (Other); Poznan University of Medical Sciences (Other); University Medical Centre Ljubljana (Other); IRCCS Burlo Garofolo (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: 36-041 ex 23/24
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neurodevelopmental Disability; Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIRS (Near-infrared spectroscopy) group of the COSGOD III trial: A multi-center, multi-national randomized-controlled trial was performed in 11 centers in Europe and Canada. Preterm neonates less than 32 weeks gestation were randomly assigned to standard care plus cerebral oxygen saturation monitoring with a dedicated treatment guideline (NIRS-group) during immediate transition (first 15 minutes after birth) and resuscitation.
  In the NIRS-group 252 (82.9%) out of 303 neonates (gestational-age, median (interquartile-range): 28.9 (26.9-30.6) weeks) survived without cerebral injury until term age or discharge. (primary outcome of the COSGOD III trial)
  Interventions: Other: NIRS group
- Control group of the COSGOD III trial: A multi-center, multi-national randomized-controlled trial was performed in 11 centers in Europe and Canada. Preterm neonates less than 32 weeks gestation were randomly assigned to standard care (control-group) during immediate transition (first 15 minutes after birth) and resuscitation.
  In the Control-group 238 (78.5%) out of 304 neonates (gestational-age, median (interquartile-range): 28.6 (26.6-30.6) weeks) survived without cerebral injury until term age or discharge. (primary outcome of the COSGOD III trial)

INTERVENTIONS:
Other: NIRS group — Standard care plus cerebral oxygen saturation monitoring with a dedicated treatment guideline (NIRS-group) during immediate transition (first 15 minutes after birth) and resuscitation.
  Groups: NIRS (Near-infrared spectroscopy) group of the COSGOD III trial

SUMMARY:
The COSGOD III trial performed follow up until term age or discharge from the neonatal intensive care unit, whatever came first. The first neonate was randomised in September 2017 and the last in October 2021. A prospective follow up of the included neonates until an age of two years was not feasible in the COSGOD III trial since funding for long-term follow-up was not available.

However, data on long-term outcome of the included neonates into COSGOD III trial are of high interest. In many centres, who participated in the COSGOD III trial neonates are assessed routinely for long term outcome in outpatient clinics with Bayleys III/IV test or PARCA-R (Parent Report of Children's Abilities) questionnaire.

Aim of the present study is therefore to analyse in neonates, who were included into the COSGOD III trial, in a retrospective observational study routinely performed long-term survival and neurodevelopmental outcome assessment at a corrected age of 2 years (18-30 months).

ELIGIBILITY:
Inclusion Criteria:

* > 50% 2 year neurodevelopmental outcome assessment at 2 years (18 to 30 months)

Exclusion Criteria:

* < 50% 2 year neurodevelopmental outcome assessment at 2 years (18 to 30 months)

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates included in COSGOD III trial
Sampling Method: Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Composite of survival without moderate to severe neurodevelopmental disability (NDD) at 2 years (18 to 30 months) corrected age | 2 years (18 to 30 months) corrected age
  A child will be classified with moderate-or-severe NDD, if any of the four following conditions are present:
  Cognitive or language disability Bayley II test cognitive scale cut-off will be < 85 Bayley III/IV test, cognitive or language composite scale cut-off will be < 85 PARCA R non-verbal cognition or language score cut-off will be < 70
  If no standardized developmental assessment is available, informal assessment is possible:
  less than 5 words
  Cerebral palsy Gross Motor Function Classification Score (GMFCS) ≥ 2
  If no GMFCS is available, informal assessment is possible:
  Not able to walk alone
  Visual impairment:
  Impairment even with glasses or only being able to perceive light or being blind (one or two eyes)
  Hearing impairment Impairment defined as hearing loss corrected with aids or being deaf

OTHER OUTCOMES:
Death | 2 years (18 to 30 months) corrected age
  Mortality mentioned in Patients charts
Conditions of neurodevelopmental outcome - Bailey Scores | 2 years (18 to 30 months) corrected age
  Testing or information from Patients charts Bailey Scores
Conditions of neurodevelopmental outcome- PARCA-R Score | 2 years (18 to 30 months) corrected age
  Testing or information from Patients charts PARCA-R Scores
Conditions of neurodevelopmental outcome - GMFC Scores | 2 years (18 to 30 months) corrected age
  Testing or information from Patients charts GMFC Scores
Weight | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Length | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Head circumference | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Long term medications | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Presence of chronic diseases | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Sex | 2 years (18 to 30 months) corrected age
  Documented in Patients charts
Gestational age | 2 years (18 to 30 months) corrected age
  Documented in Patients charts

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, Prof, Principal Investigator — Medical University of Graz
Locations (11):
- Austria (3):
  - Medical University of Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Medical University Vienna, Vienna
- University of Alberta, Edmonton, Canada
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Centre for Ped. Clinical Studies Tübingen, Tübingen
- University College Cork, Cork, Ireland
- Italy (2):
  - Ospedale dei Bambini "V.Buzzi" Milano, Milan
  - Institute for Maternal and Child Health, IRCCS Burlo Garofolo, Trieste
- Ginekologiczno Położniczy Szpital Kliniczny Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan, Poland
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pichler G, Goeral K, Hammerl M, Perme T, Dempsey EM, Springer L, Lista G, Szczapa T, Fuchs H, Karpinski L, Bua J, Avian A, Law B, Urlesberger B, Buchmayer J, Kiechl-Kohlendorfer U, Kornhauser-Cerar L, Schwarz CE, Grundler K, Stucchi I, Schwaberger B, Klebermass-Schrehof K, Schmolzer GM; COSGOD III study group. Cerebral regional tissue Oxygen Saturation to Guide Oxygen Delivery in preterm neonates during immediate transition after birth (COSGOD III): multicentre randomised phase 3 clinical trial. BMJ. 2023 Jan 24;380:e072313. doi: 10.1136/bmj-2022-072313. PMID 36693654